CLINICAL TRIAL: NCT06609720
Title: Evaluation of Autogenous Dentin Graft Versus Demineralized Freeze-Dried Bone Allograft in the Treatment of Class ΙΙ and ΙΙΙ Mandibular Furcation Defects
Brief Title: Randomized Clinical and Radiographic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Banan Lotfy Mohamed Amer, Assistant lecturer at periodontology department, Principal Investigator, MSC, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMPDR
Record Dates: First submitted 2023-12-05; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2021-02

CONDITIONS: Autogenous Dentin Graft
Keywords: dentin graft, tooth graft
MeSH Terms: interventions — Guided Tissue Regeneration

STUDY DESIGN:
Intervention Model Description: 2 groups with 2 subgroups, each subgroup receive either ADG or DFDBA
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 subgroup A (Experimental): Grade II furcation involvement treated with autogenous dentin graft
  Interventions: Procedure: (guided tissue regeneration)
- Group 1 Subgroup B (Experimental): Grade II furcation involvement treated with demineralized freeze-dried bone allograft
  Interventions: Procedure: (guided tissue regeneration)
- Group II subgroup A (Experimental): Grade III furcation involvement treated with Autogenous dentin graft
  Interventions: Procedure: (guided tissue regeneration)
- Group II subgroup B (Experimental): Grade III furcation involvement treated with demineralized freeze-dried bone allograft
  Interventions: Procedure: (guided tissue regeneration)

INTERVENTIONS:
Procedure: (guided tissue regeneration) — Randomized clinical and radiographic trial

SUMMARY:
Randomized clinical and radiographic trial

DETAILED DESCRIPTION:
Evaluation of Autogenous Dentin Graft versus Demineralized Freeze-Dried Bone Allograft in the Treatment of Class ΙΙ and ΙΙΙ Mandibular Furcation Defects

ELIGIBILITY:
Inclusion Criteria:

-

Presence of class II and/or ΙΙΙ furcation defects in mandibular first or second molars according to criteria outlined by Hamp et. al. 1975.

* Horizontal probing depth ≥3 mm using Naber's probe.
* Clinical attachment level ≥3 mm measured from cemento-enamel junction (CEJ) till the deepest probing depth.
* Evidence of radiolucency in the furcation area on panoramic radiograph.
* Patients who will be assigned for groups (I and II) should present with teeth required for extraction due to advanced periodontal bone loss or other indications such as hopeless wisdom teeth or orthodontic indications or unrestorable fractured teeth as a source for autogenous dentin graft (ADG).

Exclusion Criteria:

* Medically compromised patients and systemic conditions precluding periodontal surgery.

  * Mandibular first or second molars with root caries or endodontic treatment.
  * Smokers, diabetics, pregnant or lactating women.
  * History of chemotherapy, radiotherapy in head and/or neck region.
  * Bisphosphonate therapy.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | Measured at baseline, 6 months and 12 months
  According to Ramfjord, clinical parameter measured by UNC periodontal probe from a fixed point to the deepest probing depth. Using stent to standardize the measurements.
Clinical attachment level | Measured at baseline, 6 months and 12 months
  According to Ramfjord, clinical parameter measured by a Naber's probe. Using stent to standard measurements.
Bleeding on probing | Measured at baseline, 6 months and 12 months
  According to Ramfjord, the bleeding at each site observed after probing and recorded positive if bleeding was observed within 30 seconds, if not was recorded as negative.

SECONDARY OUTCOMES:
Radiographic outcome | measured at baseline and 1 year follow up
  Using CBCT software to analyse furcation volume

CONTACTS AND LOCATIONS:
Overall Officials: Banan L Amer, Master, Principal Investigator — Tanta University; Samia A Darwish, Professor, Study Director — Tanta University
Locations (1):
- Faculty of dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No